CLINICAL TRIAL: NCT02940223
Title: Effects of Fish Oil and Physical Activity on Fatigue in Patients With Advanced Cancer
Brief Title: Ethyl Icosapentate and Physical Activity in Treating Fatigue in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI is requesting termination (closure) of this study.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016-0348; NCI-2016-01932 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0348 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Advanced Malignant Neoplasm; Fatigue
MeSH Terms: conditions — Fatigue | interventions — eicosapentaenoic acid ethanolamide; eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (ethyl icosapentate, physical activity) (Experimental): Patients receive ethyl icosapentate PO BID for 8 weeks. Patients complete resistance exercises 3 days per week and undergo walking program at least 5 days per week for 8 weeks. After 8 weeks, patients may optionally continue to receive ethyl icosapentate, complete resistance exercises, and undergo walking program for 4 weeks.
  Interventions: Drug: Ethyl Icosapentate; Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Behavioral: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (placebo, physical activity) (Experimental): Patients receive placebo PO BID for 8 weeks. Patients complete resistance exercises 3 days per week and undergo walking program at least 5 days per week for 8 weeks. After 8 weeks, patients may optionally receive ethyl icosapentate, complete resistance exercises, and undergo walking program for 4 weeks as in Group I.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Placebo; Behavioral: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group III (placebo, stretching exercises) (Experimental): Patients receive placebo PO BID for 8 weeks. Patients meet with an exercise specialist during the first week to learn different stretching exercises and complete the stretching exercises 3 days per week for 8 weeks. After 8 weeks, patients may optionally receive ethyl icosapentate, complete resistance exercises, and undergo walking program for 4 weeks as in Group I.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Placebo; Behavioral: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Ethyl Icosapentate — Given by mouth 2 gm orally daily plus physical activity
  Other Names: ICOSAPENT ETHYL
  Arms: Group I (ethyl icosapentate, physical activity)
Behavioral: Exercise Intervention — Complete resistance exercises and undergo walking program
  Arms: Group I (ethyl icosapentate, physical activity); Group II (placebo, physical activity)
Behavioral: Exercise Intervention — Meet with exercise specialist and complete stretching exercises
  Arms: Group III (placebo, stretching exercises)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group II (placebo, physical activity); Group III (placebo, stretching exercises)
Behavioral: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well ethyl icosapentate and physical activity work in treating fatigue in patients with cancer that has spread from where it started to other places in the body. Ethyl icosapentate and physical activity may provide more robust and clinically effective improvement of cancer related fatigue, which may facilitate patients continuing cancer therapy since it would be tolerated and effective in controlling disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of the combination of ethyl icosapentate (icosapent ethyl) 2 gm orally daily plus physical activity (PA) for the reduction of cancer related fatigue (CRF) (Functional Assessment of Chronic Illness Therapy - Fatigue [FACIT-F] subscale) at the end of 8 weeks in patients with advanced cancer by comparing the difference between the FACIT-F subscale score at baseline and at 57 +/- 5 days, between patients who will receive either Icosapent ethyl plus physical activity and placebo plus physical activity.

SECONDARY OBJECTIVES:

I. To determine the feasibility, adherence, and satisfaction of using the combined intervention for the reduction of cancer related fatigue in advanced cancer.

II. To explore the effects of the combination of Icosapent ethyl 2 gm orally daily plus physical activity on quality of life (QOL)-related variables, mood (HADS - Hospital Anxiety and Depression Inventory), quality of life domains (Functional Assessment of Cancer Therapy - General [FACT-G]), cancer related symptoms (Edmonton Symptom Assessment Scale - ESAS) in these patients.

III. To explore the effects of combined intervention on serum C - reactive protein and intracellular cytokine levels (IL-6, TNF-a, IL-10, IL-1RA) before and after treatment.

IV. To explore its side effects and tolerability of the combined study interventions in these patients.

V. To explore the effect of multimodal therapy on body composition. VI. To explore the effect of the proposed treatment in this study on the overall survival time in patients.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I: Patients receive ethyl icosapentate orally (PO) twice daily (BID) for 8 weeks. Patients complete resistance exercises 3 days per week and undergo walking program at least 5 days per week for 8 weeks. After 8 weeks, patients may optionally continue to receive ethyl icosapentate, complete resistance exercises, and undergo walking program for 4 weeks.

GROUP II: Patients receive placebo PO BID for 8 weeks. Patients complete resistance exercises 3 days per week and undergo walking program at least 5 days per week for 8 weeks. After 8 weeks, patients may optionally receive ethyl icosapentate, complete resistance exercises, and undergo walking program for 4 weeks as in Group I.

GROUP III: Patients receive placebo PO BID for 8 weeks. Patients meet with an exercise specialist during the first week to learn different stretching exercises and complete the stretching exercises 3 days per week for 8 weeks. After 8 weeks, patients may optionally receive ethyl icosapentate, complete resistance exercises, and undergo walking program for 4 weeks as in Group I.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced cancer
* Patients should describe fatigue as being present for a minimum of 2 weeks
* Patients should rate the severity of fatigue as 4/10 in a 0-10 ESAS scale, where 0 = no fatigue, 10 = worse fatigue possible
* If patients are on opioids for the treatment of cancer pain, they must have had no major dose change (> 25%) for at least 48 hours prior to study entry; change in opioid dose after study entry is allowed
* Presence of relatively intact cognition defined by normal memorial delirium assessment scale (< 7/30); sign written informed consent
* Patient willing to keep a daily diary, engage in telephone follow up with a nurse
* Patient must have telephone access to be contacted by the research nurse
* Hemoglobin of >= 10 g/dl within 2 weeks of enrollment; if the patient has not had blood drawn for a hemoglobin level in the past two weeks, one will be done to determine the eligibility
* Patients should have a Zubrod =< 1
* Life expectancy of >= 4 months
* Subjects must be able to understand and be willing to sign the written informed consent form; a signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure
* Total bilirubin =< 1.5 x the upper limits of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer)
* Alkaline phosphatase limit =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer)
* Serum creatinine =< 1.5 x the ULN
* International normalized ratio (INR)/ partial thromboplastin time (PTT) =< 1.5 x ULN
* Platelet count > 100000/mm^3
* Hemoglobin (Hb) > 9 g/dL
* Absolute neutrophil count (ANC) 1500/mm^3
* Blood transfusion to meet the inclusion criteria will not be allowed
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug; post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test; the definition of adequate contraception will be based on the judgment of the investigator
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent form (ICF) until at least 2 months after the last dose of study drug; the definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate
* Subject must be able to swallow and retain oral medication
* Patients on pain medications (non-opioids), including nonsteroidal anti-inflammatory drugs (NSAIDS) and acetaminophen, may be enrolled as long as they have been using it chronically, at least more than 2 weeks

Exclusion Criteria:

* Major contraindication to fish oil i.e. hypersensitivity to fish/oil or physical activity
* Currently on fish oil or has been on fish oil within the last 10 days
* Inability to complete the baseline assessment forms or to understand the recommendations for participation in the study
* Pregnant or lactating women; childbearing age women are not on birth control
* Reports a fall in the past 30 days
* Patient reported regular participation in moderate- or vigorous-intensity physical activity for at >= 30 minutes at least 5 times a week and strength training for >= 2 days/week
* Signs of third spacing as determined by the treating physician (e.g., pedal edema, pleural effusion, ascites)
* Previous assignment to treatment during this study; subjects permanently withdrawn from study participation will not be allowed to re-enter study
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0] on repeated measurement) despite optimal medical management
* Active or clinically significant cardiac disease including: a. congestive heart failure-New York Heart Association (NYHA) > class II; b. active coronary artery disease; c. cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin; d. unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization
* Evidence or history of bleeding diathesis or coagulopathy
* Any hemorrhage or bleeding event >= NCI CTCAE grade 3 within 4 weeks prior to start of study medication
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of study treatment within 6 months of informed consent
* Patients with any previously untreated or concurrent cancer that is distinct in primary site or histology except cervical cancer in-situ, treated ductal carcinoma in situ of the breast, curatively treated nonmelanoma skin carcinoma, noninvasive aerodigestive neoplasms, or superficial bladder tumor; subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before registration are allowed; all cancer treatments must be completed at least 3 years prior to registration
* Patients with phaeochromocytoma
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy
* Ongoing infection > grade 2 NCI-CTCAE v4.0
* Symptomatic metastatic brain or meningeal tumors
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* Major surgical procedure or significant traumatic injury within 28 days before start of study medication
* Renal failure requiring hemo-or peritoneal dialysis
* Dehydration grade > 1 NCI-CTCAE v4.0
* Patients with seizure disorder requiring medication
* History of persistent proteinuria >= grade 3 NCI-CTCAE v4.0
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Pleural effusion or ascites that causes respiratory compromise (>= NCI-CTCAE version 4.0 grade 2 dyspnea); a) history of organ allograft (including corneal transplant); b) known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial; c) any malabsorption condition; d) any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation; e) substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 4 weeks of trial entry (signing of the informed consent form)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication
* Therapeutic anticoagulation with vitamin-K antagonists (e.g., warfarin) or with heparins and heparinoids; however, prophylactic anticoagulation as described below is allowed: 1. low dose warfarin (1 mg orally, once daily) with prothrombin time [PT]-INR =< 1.5 x ULN is permitted; we will monitor the PT/INR weekly for patients on warfarin and liver function test every 2 weeks (total bilirubin, and AST (serum glutamic oxaloacetic transaminase [SGOT]) and ALT (serum glutamic pyruvic transaminase [SGPT]) if hepatic metastases are present or if patients are on potentially hepatoxic agents such as acetaminophen or statins; 2. low dose aspirin (=< 100 mg daily); and 3. prophylactic doses of heparin
* Use of any herbal remedy (e.g. St. John's wort [Hypericum perforatum])
* Use of dexamethasone for cancer related fatigue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with advanced cancers aged >=18 years with fatigue for 2 weeks were recruited from MD Anderson Cancer Center between 3/16/2017 (check activation date) and 10/2/2017 (check last patient off study date).
Pre-assignment Details: A total of 2 participants were recruited before the study was aborted due to low accrual..
Groups:
- Intervention Group (Icosapent Ethyl): Received 1 mg Icosapent Ethyl capsules orally twice a daily plus physical activity for 8 weeks
- Placebo: Received placebo capsules orally twice a day plus physical activity for 8 weeks
Period: Overall Study
Arm/Group | Intervention Group (Icosapent Ethyl) | Placebo
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Failed Requirement | 2 | 0

BASELINE CHARACTERISTICS:
Population: A total of 2 participants were recruited before the study was aborted due to low accrual.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Icosapent Ethyl) | Placebo | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2
Cancer Type [Count of Participants; unit: Participants]
  Colorectal | 1 | 0 | 1
  Hepatic | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cancer Related Fatigue
Description: Cancer related fatigue was measured using the 13 questions of Functional Assessment of Chronic Illness Therapy - Fatigue subscale on a four point Likert scale (0=not at all fatigue to 4= very much fatigued). We measured the difference in Functional Assessment of Chronic Illness Therapy - Fatigue subscale score between baseline and 57±5 days, among patients who would receive either Icosapent ethyl plus physical activity and placebo plus physical activity.
Time Frame: Baseline and at 57±5 days
Population: Due to low accrual and early termination of the protocol no analysis was done to determine the Cancer related fatigue.
Arm/Group | Intervention Group (Icosapent Ethyl) | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Edmonton Symptom Assessment System (ESAS) Score
Description: Edmonton Symptom Assessment System score was measured using 10 question Edmonton Symptom Assessment System form with 0-10 scale with 0= no symptom and 10=worst symptom imaginable. We measured the difference in Edmonton Symptom Assessment System score between baseline and 57±5 days, among patients who would receive either Icosapent ethyl plus physical activity and placebo plus physical activity.
Time Frame: Baseline and at 57±5 days
Population: Due to low accrual and early termination of the protocol no analysis was done to determine the Edmonton Symptom Assessment System score.
Arm/Group | Intervention Group (Icosapent Ethyl) | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Hospital Anxiety and Depression Score
Description: Hospital Anxiety and Depression score was measured using 14 questions HADS form with 0-4 scale with 0= no symptom and 4=worst symptom. We measured the difference in Hospital Anxiety and Depression score between baseline and 57±5 days, among patients who would receive either Icosapent ethyl plus physical activity and placebo plus physical activity.
Time Frame: Baseline and at 57±5 days
Population: Due to low accrual and early termination of the protocol no analysis was done to determine the Hospital Anxiety and Depression score.
Arm/Group | Intervention Group (Icosapent Ethyl) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Description: Due to low accrual and early termination of the protocol there were no adverse events collected.
Arm/Group | Intervention Group (Icosapent Ethyl) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT02940223/Prot_SAP_000.pdf